CLINICAL TRIAL: NCT06098170
Title: Acceptance and Commitment Therapy for Chronic Pain in SCI: Development and Testing of an eHealth Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Anna Kratz, Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00192610
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injuries
Keywords: My SCI Toolkit; eHealth-delivered Acceptance and Commitment Therapy (ACT) intervention; Chronic pain
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled and randomized 1:1:1 to receive unguided use of the My SCI Toolkit program (number (n)=20), coached My SCI Toolkit (n=20) or wait-list control (n=20; treatment as usual) for an 8-week treatment period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unguided use of the My SCI Toolkit program (Experimental)
  Interventions: Behavioral: Unguided use of the My SCI Toolkit program
- Coached My SCI Toolkit (Experimental)
  Interventions: Behavioral: Coached My SCI Toolkit
- Wait-list control (No Intervention): Participants will not access the My SCI Toolkit program during the 8-week study period and will be asked to continue daily life, including management of pain, as usual.

INTERVENTIONS:
Behavioral: Unguided use of the My SCI Toolkit program — Participants will be asked to use the My SCI Toolkit program for 8 weeks (without a coach), following the prompts and guides built into the program.
  Arms: Unguided use of the My SCI Toolkit program
Behavioral: Coached My SCI Toolkit — Participants will be asked to use the My SCI Toolkit program for 8 weeks, following the prompts and guides built into the program. Participants will also have weekly phone calls (the first is about 30-45 minutes, and the rest are about 15 minutes) with a study coach. The coach can help answer questions and tailor the skills more to the participant's goals and needs. The coaching sessions will be audio recording for fidelity purposes.
  Arms: Coached My SCI Toolkit

SUMMARY:
This study will test the newly-developed My spinal cord injury (SCI) Toolkit program in two formats - unguided use of the program and use supported by a coach. These two active treatment formats will be compared to treatment as usual (waitlist control) in adults with chronic pain and SCI.

Hypotheses include:

* Treatment adherence, participant satisfaction, and perception of positive change will be high and drop-out rates low for both treatments but will be better in the coached compared to the unguided arm
* In terms of pre- to post-treatment changes in pain interference, coached My SCI Toolkit program will be superior to treatment as usual

DETAILED DESCRIPTION:
All participants will also be asked to complete online surveys at baseline (before being randomized to a group), half-way through the 8-week study period, and after the 8-week study period is over. The surveys are online and can be completed from home. Participants in the unguided and coached programs will also be asked to complete a weekly online survey asking about use of the website in the past week, taking approximately 5 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCI (all injury levels included);
* Average pain intensity over the past 3 months greater or equal to (≥) 4/10 on 0-10 numerical rating scale
* Fluent in English and able to read English at a 6th grade level
* Access to internet connected device (phone, tablet, computer) and telephone
* Willingness to maintain stable analgesic regimen during study period

Exclusion Criteria:

* Currently in inpatient care or intensive outpatient physical therapy
* Significant cognitive impairment as indicated by scores ≥2 on cognitive screener

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-07-21 (Actual)

PRIMARY OUTCOMES:
Percent of participants in each arm that dropped out of the study | 8 weeks
Number of days/week that My SCI Toolkit was accessed | 8 weeks
Number of minutes/week spent on the My SCI Toolkit website | 8 weeks
Participant Satisfaction Evaluation | 8 weeks (post intervention)
  This is a 12-question survey that participants answer with scores ranging from 1-4. The total scores range from 12-48 with a higher score meaning more satisfaction.
Patient Global Impression of Change (PGIC) | 8 weeks (post intervention)
  This is a one question scale that participants select from no change (1) to a great deal better (7).
Change in SCI-QOL Pain Interference Short Form | Baseline, 8 weeks (post intervention)
  This is a 10-question survey that participants answer from not at all (1) to very much (5).
  Scores are on a T-score metric with Mean=50, Standard Deviation=10. A higher score means more interference.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Short Form | Baseline, 8 weeks (post intervention)
  This is a 3-question survey that is scored on a T-score metric with Mean=50, Standard Deviation=10. A higher score means higher pain intensity.
Change in SCI-QOL Pain Behavior Short Form | Baseline, 8 weeks (post intervention)
  This survey has 7-questions. Three questions are answered never (1) to always (5) and 3 questions are answered had no pain (1) to always (6). Scores are on a T-score metric with a Mean=50, Standard Deviation=10. A higher score indicates more behavioral manifestations of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kratz, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT06098170/ICF_000.pdf